CLINICAL TRIAL: NCT02933242
Title: Phase II Non-randomized Trial of Stereotactic Ablative Radiotherapy (SABR) for Oligometastases
Brief Title: Stereotactic Ablative Body Radiotherapy (SABR) for Oligometastases
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Principal Investigator, Robert Olson, Radiation Oncologist, British Columbia Cancer Agency
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H16-02233
Record Dates: First submitted 2016-10-06; First posted 2016-10-14 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Tumors
Keywords: Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic arm (Experimental): Stereotactic ablative radiotherapy
  Interventions: Radiation: Stereotactic Ablative Body Radiotherapy

INTERVENTIONS:
Radiation: Stereotactic Ablative Body Radiotherapy — The total dose and number of fractions will depend on the site of disease. Treatment will be given daily, or every other day, over 1 -3 weeks
  Other Names: SABR; SBRT

SUMMARY:
This is a study measuring toxicity while making observations about the survival benefits of treating participants with oligometastatic disease using stereotactic ablative radiotherapy (SABR).

DETAILED DESCRIPTION:
To assess quality of life and side effects in participants with up to 5 metastatic cancer lesions treated with a comprehensive oligometastatic SABR treatment program. Secondarily, the investigators will document the disease free and overall survival.

Rationale:

The oligometastatic state was first defined in 1995 and refers to a stage of disease where cancer has spread beyond the site of origin, but is not yet widely metastatic. In such a state of limited metastatic disease, it is hypothesized that eradication of all sites of metastatic disease could result in long-term survival, or even cure, in some participants. Ablation of metastatic deposits can be achieved through several techniques, including surgery, radiofrequency ablation (RFA), or through Stereotactic ablative body radiotherapy (SABR), a new radiotherapy technology that delivers very large, hypofractionated doses of radiotherapy to small tumor targets, with high rates of local control.

Clinical evidence to support the presence of an oligometastatic state is controversial. However, there is emerging low quality evidence in both the surgical and SABR literature that this state may exist. In a study of over 5200 participants with lung metastases who underwent surgical resection, a 5-year survival of 36% was reported in participants who achieved a complete resection, much higher than would be expected for stage IV disease.3 Similarly, in participants treated with SABR for 1-3 lung metastases from a variety of primary tumors, local control with SABR was 96% at 2-years, and 2-year survival was 39%. Long-term survival has been demonstrated in participants treated for oligometastases with surgery or SABR at several other tumor sites, including liver, brain, bone, and adrenal metastases. The risk of further metastases after ablative treatment is up to 60-80% in some studies. SABR can also be used for further salvage at newly progressive sites (oligoprogression).

Despite the apparent achievement of long-term survival with ablative treatment for oligometastatic disease, the level of evidence to support such treatments is weak, often based on single-arm studies without appropriate controls. Participants included in such reports are highly selected, based on good performance status and slow pace of tumor progression. It has been suggested that the long-term survival achieved with treatment of oligometastases is a result of the selection of fit participants with very slow-growing tumors, rather than the result of treatment intervention.

Randomized trials are therefore necessary to establish the utility of ablative treatment of oligometastatic disease, and therefore the BCCA oligometastatic SABR group, recommends that participants be considered for a randomized control before being offered SABR on this current trial. In some circumstances, participants may not be comfortable with this approach, or their physicians do not have clinical equipoise, and therefore SABR for oligometastatic disease may be appropriate. BCCA has decided that given the limited evidence for SABR in this setting, it will not be offered off trial. The main focus of this trial is to assess the side effects and quality of life post SABR. This trial aims to provide a clear informed consent process, including the limited evidence for SABR off trial, and potential harm from SABR, for participants opting to pursue SABR for oligometastases.

This is a non-randomized phase II trial where all participants will receive experimental SABR to all sites of metastatic disease. The investigators will accrue 200 participants to assess toxicity associated with this experimental treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Histologically confirmed malignancy with metastatic disease detected on imaging.

  * Biopsy of metastasis is preferred, but not required.
* Primary tumour treated radically or controlled by prior palliative radiotherapy or systemic therapy
* Maximum 5 metastases eligible for SABR (either 5 in total or 5 not controlled by prior treatment)
* Standard of care tests prior to SABR CT simulation within 14 weeks:

  * Brain CT or MRI imaging (for tumour sites with propensity for brain metastasis)
  * Body imaging:
* CT chest/abdomen/pelvis, with or without bone scan (at discretion of study doctor), required if no PET-CT is performed
* PET-CT or PSMA-PET is only required for specific evidence-based indications, and in such cases the CT neck/chest/abdomen/pelvis and bone scan are not required:
* MRI spine for patients with vertebral or paraspinal metastases

  * For other indications, at the discretion of the treating oncologists, e.g. PET-CT scans may be done but are not required.
  * Blood tests as per standard of care
  * Pregnancy test for women of child-bearing age
* ECOG performance status 0-2
* All sites of progressive disease can be safely treated based on criteria below
* For non-brainstem mets, maximum size of 3cm if using single fraction radiosurgery.

  * If size is from 3.1 to 4cm, 25-35Gy/5 can be considered
* All brain metastases cases need approval from Stereotactic Radiosurgery (SRS) rounds

  * Maximum size of 6 cm for lesions outside the brain, except:
* Bone metastases over 6 cm may be included, if in the opinion of the local PI it can be treated safely (e.g. rib, scapula, pelvis)
* Life expectancy > 6 months

  * In many scenarios, this is best estimated by a multidisciplinary opinion from disease site experts, often obtained by presentation at multidisciplinary tumours rounds.
* Not a candidate for surgical resection at all sites: surgery to all sites not recommended by multidisciplinary team, or unfit or declining surgery.
* No chemotherapy agents (cytotoxic, or molecularly targeted agents) will be used within the period of time commencing 2 weeks prior to radiation, lasting until 1 week after the last fraction. Certain chemotherapy agents may require a longer break prior to or after SABR if protocols dictate. Hormonal therapy during SABR is allowed.
* Patients with metastases that have been previously treated may be eligible for this SABR protocol:

  * If the previous treatment was systemic therapy, the patient may be eligible, if the metastases have demonstrated a complete radiologic response
  * If the previous treatment was by a local non-radiation means (e.g. prior resection, RFA or microwave ablation), then SABR may be considered for residual/recurrent disease
  * If the previous treatment was SABR, the patient is not eligible unless the new site(s) was/were not previously treated
* If the previous treatment was conventional RT, SABR could be considered if it can be delivered safely. In such a circumstance it must be presented in a multidisciplinary setting for approval.
* Review and consensus by 3 disease site experts, or tumour group conference, for eligibility/prognosis Patients must be able and willing to complete quality of life questionnaires in English, and other assessments that are a part of this study, via paper or online using REDCap (if email address is provided by participant on the informed consent) Note: The potential treating SABR radiation oncologist reserves the right to require a multidisciplinary note documenting life expectancy, other treatment options and suitability for SABR.

Exclusion Criteria:

* Serious medical co-morbidities precluding radiotherapy
* Bone metastasis in a femoral bone if risk of pending fracture is high
* Participants with 1-3 brain metastasis and no disease elsewhere (these participants should not be accrued but treated with stereotactic radiotherapy as per results of published randomized trials)
* Complete response to first-line chemotherapy (i.e. no measurable target for SABR)
* Persistent malignant pleural effusion
* Inability to treat all sites of active disease with ablative intent
* Clinical or radiological evidence of spinal cord compression
* Dominant brain metastasis requiring surgical decompression
* a candidate for a clinical trial that randomizes between SABR and a standard treatment
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2016-11; Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Patient-reported Quality of life, function and health status using BC Cancer's Prospective Outcomes and Support Initiative (POSI). | At approximately end of year 5 (end of study)
  Measuring percentage change in patient reported QoL before and after SABR treatment
Toxicity as Assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4 for each organ treated (e.g. liver, lung, bone)] | At approximately the end of year 1
  Prevalence of various SAE graded events
Toxicity as Assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4 for each organ treated (e.g. liver, lung, bone)] | At approximately the end of year 2
  Prevalence of various SAE graded events
Toxicity as Assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4 for each organ treated (e.g. liver, lung, bone)] | At approximately the end of year 3
  Prevalence of various SAE graded events
Toxicity as Assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4 for each organ treated (e.g. liver, lung, bone)] | At approximately the end of year 4
  Prevalence of various SAE graded events
Toxicity as Assessed by the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 4 for each organ treated (e.g. liver, lung, bone)] | At approximately the end of year 5
  Prevalence of various SAE graded events

SECONDARY OUTCOMES:
Overall survival | At approximately end of year 5 (end of study)
  Defined as time until death from any cause
Progression-free survival | At approximately end of year 5 (end of study)
  Defined as time to either progression or death
Lesional control rate, defined as lack of further progression | At approximately end of year 5 (end of study)
  Assessed retrospectively using RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Robert Olson, MD, Principal Investigator — BC Cancer Agency - Centre for the North
Locations (1):
- BC Cancer, Prince George, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louie AV, Rodrigues G, Yaremko B, Yu E, Dar AR, Dingle B, Vincent M, Sanatani M, Younus J, Malthaner R, Inculet R. Management and prognosis in synchronous solitary resected brain metastasis from non-small-cell lung cancer. Clin Lung Cancer. 2009 May;10(3):174-9. doi: 10.3816/CLC.2009.n.024. PMID 19443337
- [Background] Milano MT, Katz AW, Schell MC, Philip A, Okunieff P. Descriptive analysis of oligometastatic lesions treated with curative-intent stereotactic body radiotherapy. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1516-22. doi: 10.1016/j.ijrobp.2008.03.044. Epub 2008 May 19. PMID 18495378
- [Background] Inoue T, Katoh N, Aoyama H, Onimaru R, Taguchi H, Onodera S, Yamaguchi S, Shirato H. Clinical outcomes of stereotactic brain and/or body radiotherapy for patients with oligometastatic lesions. Jpn J Clin Oncol. 2010 Aug;40(8):788-94. doi: 10.1093/jjco/hyq044. Epub 2010 Apr 20. PMID 20406944
- [Background] Milano MT, Philip A, Okunieff P. Analysis of patients with oligometastases undergoing two or more curative-intent stereotactic radiotherapy courses. Int J Radiat Oncol Biol Phys. 2009 Mar 1;73(3):832-7. doi: 10.1016/j.ijrobp.2008.04.073. Epub 2008 Aug 28. PMID 18760543
- [Background] Treasure T, Fallowfield L, Farewell V, Ferry D, Lees B, Leonard P, Macbeth F, Utley M; Pulmonary Metastasectomy in Colorectal Cancer (PulMiCC) trial development group. Pulmonary metastasectomy in colorectal cancer: time for a trial. Eur J Surg Oncol. 2009 Jul;35(7):686-9. doi: 10.1016/j.ejso.2008.12.005. Epub 2009 Jan 18. PMID 19153025
- [Background] Primrose J, Treasure T, Fiorentino F. Lung metastasectomy in colorectal cancer: is this surgery effective in prolonging life? Respirology. 2010 Jul;15(5):742-6. doi: 10.1111/j.1440-1843.2010.01759.x. Epub 2010 Apr 23. PMID 20456671
- [Background] Timmerman RD. An overview of hypofractionation and introduction to this issue of seminars in radiation oncology. Semin Radiat Oncol. 2008 Oct;18(4):215-22. doi: 10.1016/j.semradonc.2008.04.001. No abstract available. PMID 18725106
- [Result] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Result] Macdermed DM, Weichselbaum RR, Salama JK. A rationale for the targeted treatment of oligometastases with radiotherapy. J Surg Oncol. 2008 Sep 1;98(3):202-6. doi: 10.1002/jso.21102. PMID 18618604
- [Result] Pastorino U, Buyse M, Friedel G, Ginsberg RJ, Girard P, Goldstraw P, Johnston M, McCormack P, Pass H, Putnam JB Jr; International Registry of Lung Metastases. Long-term results of lung metastasectomy: prognostic analyses based on 5206 cases. J Thorac Cardiovasc Surg. 1997 Jan;113(1):37-49. doi: 10.1016/s0022-5223(97)70397-0. PMID 9011700
- [Result] Rusthoven KE, Kavanagh BD, Burri SH, Chen C, Cardenes H, Chidel MA, Pugh TJ, Kane M, Gaspar LE, Schefter TE. Multi-institutional phase I/II trial of stereotactic body radiation therapy for lung metastases. J Clin Oncol. 2009 Apr 1;27(10):1579-84. doi: 10.1200/JCO.2008.19.6386. Epub 2009 Mar 2. PMID 19255320
- [Result] Rusthoven KE, Kavanagh BD, Cardenes H, Stieber VW, Burri SH, Feigenberg SJ, Chidel MA, Pugh TJ, Franklin W, Kane M, Gaspar LE, Schefter TE. Multi-institutional phase I/II trial of stereotactic body radiation therapy for liver metastases. J Clin Oncol. 2009 Apr 1;27(10):1572-8. doi: 10.1200/JCO.2008.19.6329. Epub 2009 Mar 2. PMID 19255321
- [Derived] Olson R, Jiang W, Liu M, Bergman A, Schellenberg D, Mou B, Alexander A, Carolan H, Hsu F, Miller S, Atrchian S, Chan E, Ho C, Mohamed I, Lin A, Berrang T, Bang A, Chng N, Matthews Q, Baker S, Huang V, Mestrovic A, Hyde D, Lund C, Pai H, Valev B, Lefresene S, Tyldesley S. Treatment With Stereotactic Ablative Radiotherapy for Up to 5 Oligometastases in Patients With Cancer: Primary Toxic Effect Results of the Nonrandomized Phase 2 SABR-5 Clinical Trial. JAMA Oncol. 2022 Nov 1;8(11):1644-1650. doi: 10.1001/jamaoncol.2022.4394. PMID 36173619
- [Derived] Olson R, Liu M, Bergman A, Lam S, Hsu F, Mou B, Berrang T, Mestrovic A, Chng N, Hyde D, Matthews Q, Lund C, Glick D, Pai H, Basran P, Carolan H, Valev B, Lefresene S, Tyldesley S, Schellenberg D. Population-based phase II trial of stereotactic ablative radiotherapy (SABR) for up to 5 oligometastases: SABR-5. BMC Cancer. 2018 Oct 4;18(1):954. doi: 10.1186/s12885-018-4859-7. PMID 30286739

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT02933242/Prot_SAP_002.pdf
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT02933242/ICF_003.pdf